CLINICAL TRIAL: NCT03698201
Title: Are Gliomas in Adults Associated With a Unique Identifying Blood Biomarker Signature?
Brief Title: Blood Biomarker Signature in Glioma
Status: Terminated | Type: Observational
Why Stopped: As per the HRBs new funding model, HRBs investment will not support costs associated with routine patient care or translational studies, biobanks, patient registries and questionnaires. Therefore, a decision was made to cease further study follow up.
Sponsor: Cancer Trials Ireland (Network)
Collaborators: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: CTRIAL-IE (ICORG) 08-13
Record Dates: First submitted 2018-09-12; First posted 2018-10-05 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Glioma of Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 / High grade Glioma: Cohort 1:
  1. Histologically confirmed high grade glioma (grade III) or glioblastoma (GBM, astrocytoma grade IV)
  2. Planned treatment (RT alone or Chemotherapy alone or a combination of RT/Chemotherapy)
  Interventions: Other: Non-interventional
- Cohort 2 / Low grade Glioma: Cohort 2:
  1. Histologically confirmed low grade (grade II) glioma
  2. Planned treatment either
     * expectant monitoring or
     * RT alone or
     * Chemotherapy alone or
     * a combination of RT/Chemotherapy
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Translational, observational study

SUMMARY:
This is an exploratory, translational and non-interventional clinical study. The aim of this study is to identify a blood biomarker signature for glioma.

DETAILED DESCRIPTION:
The identification of biomarkers (proteins, peptides and micro RNAs (miRNAs)) in the serum of patients with glioma would be a new, less invasive approach, which could help in the diagnosis of a glioma, and potentially help guide therapeutic decisions.

The investigators will investigate the existence of biomarker profiles, which can

* distinguish between low and high grade gliomas
* correlate with patient outcomes including response to treatment and survival
* indicate progression from a low to a high grade glioma.

In this study the investigators collect and analyse blood samples taken from patients with suspected newly diagnosed grade II/III glioma or glioblastoma multiforme (GBM). Blood samples will be collected before any surgical intervention (resection or biopsy) and at various follow-up time points until progression or death. Based on the known natural history of gliomas (described above), it is planned to follow patients with grade III/IV tumours, who receive treatment, for up to 3 years and those with grade II-III tumours, (irrespective of treatment) for up to 5 years. Ultimately, the investigators envisage the translation of our observations into the hospital setting to aid the distinction between glioma grade II and grade III/IV.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with suspected newly diagnosed glioma (grade 2 or 3 or glioblastoma) with planned surgical intervention (resection or biopsy).
2. Patient aged 18 years or older
3. Patients have to be able to give informed consent

Exclusion Criteria:

1. Prior Radiotherapy to the central nervous system
2. Prior Chemotherapy within the last 5 years
3. Any prior central nervous system malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with suspected newly diagnosed glioma with planned surgical intervention will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Identification of protein and miRNA biomarker ignatures | 5 years
  Identification of protein and miRNA biomarker signatures in serum of glioma patients as assessed by surface-enhanced laser desorption ionization - time of flight (SELDI-TOF), Isobaric tags for relative and absolute quantitation (iTRAQ) and miRNA array technologies.
  Profiling experiments will be performed on the serum samples
  * to find unique glioma associated serum biomarkers
  * to determine if the levels of discovered biomarkers accurately reflect glioma grade.
  * to investigate if alterations in levels of glioma associated markers predict glioma progression from low grade to high grade Profiling patient's protein and miRNA biomarker signatures will allow association of expression patterns with tumour grade. We will determine if alterations in levels of identified serum biomarkers correlate with disease progression and patient outcome, including tumour response, time to progression (TTP) and overall survival (OS).

SECONDARY OUTCOMES:
Correlation with disease progression | 5 years
  The secondary objectives are to determine if alterations in levels of identified serum biomarkers correlate with disease progression and patient outcome, including tumour response, time to progression (TTP) and overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Prehn, Principal Investigator — Cancer Trials Ireland
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No